CLINICAL TRIAL: NCT00040859
Title: A Phase II Study of Oxaliplatin and Capecitabine in Patients With Measurable Metastatic Adenocarcinoma of the Esophagus, Gastroesophageal Junction, and Gastric Cardia
Brief Title: Oxaliplatin and Capecitabine in Treating Patients With Advanced Esophageal Cancer or Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0149; NCI-2012-02471 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000069413 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage IV gastric cancer; recurrent gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- oxaliplatin + capecitabine (Experimental): Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) receive 2 additional courses after CR.
  Quality of life is assessed at baseline and then every 3 weeks (prior to each course of chemotherapy).
  Patients are followed every 3 months for 1 year and then every 6 months for 2 years.
  Interventions: Drug: capecitabine; Drug: oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining oxaliplatin with capecitabine in treating patients who have advanced esophageal cancer or stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective tumor response rate of patients with advanced adenocarcinoma of the esophagus, gastroesophageal junction, or gastric cardia treated with oxaliplatin and capecitabine.

Secondary

* Determine the time to progression and overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen in these patients.
* Assess the quality of life of patients treated with this regimen.

OUTLINE: Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-14. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with complete response (CR) receive 2 additional courses after CR.

Quality of life is assessed at baseline and then every 3 weeks (prior to each course of chemotherapy).

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the esophagus, gastroesophageal junction, or gastric cardia for which no potentially curative or significant palliative therapy exists

  * Unresectable disease
  * Gastric cardia is defined as no more than 5 cm from the gastroesophageal junction into the stomach
* Measurable disease
* No known CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than upper limit of normal (ULN)
* AST no greater than 3 times ULN
* Alkaline phosphatase no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.5 times ULN
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Able to swallow capecitabine
* No unresolved gastrointestinal bleeding
* No uncontrolled infection
* No chronic debilitating disease
* No peripheral neuropathy grade 2 or greater
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or adequately treated noninvasive carcinoma
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy or biological therapy for recurrent or metastatic disease
* No concurrent biologic agents

Chemotherapy:

* No prior chemotherapy for recurrent or metastatic disease
* Prior adjuvant or neoadjuvant chemotherapy (including combination chemotherapy and radiotherapy) allowed
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Chemotherapy
* No prior radiotherapy for recurrent or metastatic disease
* No prior radiotherapy to more than 25% of the bone marrow
* Prior adjuvant or neoadjuvant radiotherapy allowed
* More than 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* More than 4 weeks since prior abdominal exploration with surgical resection
* More than 3 weeks since prior abdominal exploration without surgical resection

Other:

* No concurrent oral cryotherapy during oxaliplatin administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-09; Primary Completion 2005-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Objective tumor response rate | Up to 3 years

SECONDARY OUTCOMES:
Time to progression | Up to 3 years
Overall survival | Up to 3 years
Quality of life | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (6):
- United States (6):
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota

REFERENCES:
- [Background] Jatoi A, Foster NR, Egner JR, Burch PA, Stella PJ, Rubin J, Dakhil SR, Sargent DJ, Murphy BR, Alberts SR. Older versus younger patients with metastatic adenocarcinoma of the esophagus, gastroesophageal junction, and stomach: a pooled analysis of eight consecutive North Central Cancer Treatment Group (NCCTG) trials. Int J Oncol. 2010 Mar;36(3):601-6. doi: 10.3892/ijo_00000535. PMID 20126980
- [Result] Jatoi A, Murphy BR, Foster NR, Nikcevich DA, Alberts SR, Knost JA, Fitch TR, Rowland KM Jr; North Central Cancer Treatment Group. Oxaliplatin and capecitabine in patients with metastatic adenocarcinoma of the esophagus, gastroesophageal junction and gastric cardia: a phase II study from the North Central Cancer Treatment Group. Ann Oncol. 2006 Jan;17(1):29-34. doi: 10.1093/annonc/mdj063. Epub 2005 Nov 22. PMID 16303863